CLINICAL TRIAL: NCT02558491
Title: Feasibility of a Decision Support System to Reduce Glucose Variability in Subject With T1DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Chernavvsky, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Daniel Chernavvsky, MD, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18348; 5R01DK051562-18 (NIH); G150172 (Other: FDA)
Record Dates: First submitted 2015-09-02; First posted 2015-09-24 (Estimated); Results first posted 2023-03-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1DM); Artificial Pancreas Project (APP); Diabetes Assistant (DiAs); Insulin Pump; Continuous Glucose Monitor; Exercise; Glucose Variability; Decision Support System; Multiple Daily Injections (MDI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Support System (Experimental): Blinded continuous glucose monitor (CGM) data will be collected prior to the Experimental Admission and analyzed by the study team to determine the optimal insulin therapy parameters for each insulin pump and multiple daily injections (MDI) participant. These optimized parameters will be used during the Experimental Admission.
  Interventions: Device: Decision Support System
- Usual Care (Active Comparator): Insulin pump and MDI participants will use their own insulin parameters, including basal rate, correction factor and carbohydrate-insulin ratio, and determine their own insulin usage during the Control Admission.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Decision Support System — The purpose of this study is to demonstrate the safety and feasibility of a Decision Support System aimed at reducing glucose variability in T1DM patient using an insulin pump or MDI. The system will be deployed on our portable medical application platform (DiAs) and will include the following elements:
  1. An insulin pump treatment parameters optimization routine, using a month of collected CGM/insulin/meal data
  2. An exercise risk warning system, capable of predicting hypoglycemia at the onset of physical activity and advising on mitigating alteration of treatment.
  3. A smart bolus calculator based on CGM glucose measurements and insulin sensitivity estimation.
  Arms: Decision Support System
Other: Usual Care — During the Control study admission, DiAs will be programmed with the home insulin dosing parameters. The study subject will use the home basal/bolus MDI or continuous subcutaneous insulin infusion (CSII) insulin regimen via the home insulin pens or pump and determine the amount of insulin to give for the entire admission per the subject's home carb counting parameters and as calculated by the DiAs meal screen.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to demonstrate the safety and feasibility of a decision support system aimed at reducing glucose variability in T1DM patient using an insulin pump.

DETAILED DESCRIPTION:
The overall aim of this proposed research is to demonstrate the safety and feasibility of a decision support system aimed at reducing glucose variability in T1DM patient using an insulin pump. The system will be deployed on our portable medical application platform (DiAs) and will include insulin pump treatment parameters optimization and an exercise risk warning system, capable of predicting hypoglycemia at the onset of physical activity and advising on mitigating alteration of treatment.

A second phase of the trial will enroll additional users of insulin pumps, and subjects who treat their T1DM with the use of multiple daily injections (MDI) of insulin. MDI users should be administering the Lantus (glargine) dose at approximately the same time each day and use only one basal rate per day. MDI users will also use MySugr app to count carbohydrates for all meals that require insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis based on investigator assessment, of type 1 diabetes for at least one year and either using insulin pump therapy for at least 6 months or MDI therapy (consisting of a of Lantus [glargine], Tresiba [degludec], or Levemir [Detemir] plus rapid-acting meal insulin) for at least 6 months; 1-2 basal insulin injections per day, consistent in timing and amount.

   A. Historical criteria for documented hyperglycemia (at least 1 must be met):

   i. Fasting glucose ≥126 mg/dL. ii. Two-hour oral glucose tolerance test (OGTT) glucose ≥200 mg/dL. iii. Hemoglobin A1c ≥6.5% documented. iv. Random glucose ≥200 mg/dL with symptoms. v. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes.

   B. Historical criteria for requiring insulin at diagnosis (1 must be met):

   i. Participant required insulin at diagnosis and continually thereafter. ii. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually.

   iii. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually.
2. Age 21- 65years old.
3. Females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while participating in the study. A negative urine/blood pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.
4. Demonstration of proper mental status and cognition for the study
5. MDI subjects should be administering the Lantus (glargine), Tresiba [degludec], or Levemir [Detemir] dose at approximately the same time each day.
6. CSII subjects must currently be using the bolus calculator function of the current insulin pump with pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor.
7. MDI users must currently be using Intensive Insulin Therapy including carbohydrate counting and use of pre-defined parameters for glucose goal, carbohydrate ratio, and insulin sensitivity factor.
8. Willing to use Humalog (lispro) or Novolog (aspart) insulin during the study procedures for MDI subjects.
9. CSII subjects must be willing to use the current bolus calculator pump parameters and enter all carbohydrate intake into the pump during the 28 day data collection period.
10. MDI users must be willing to use their carbohydrate counting parameters for all meal dosing and enter the information into the MySugr app.
11. Ability to access the Internet to provide data to the clinical team or to travel to the research center so that the study equipment and personal pump can be downloaded.
12. An understanding of and willingness to follow the protocol and sign the informed consent.

Exclusion Criteria: The presence of any of the following is an exclusion for the study:

1. Diabetic ketoacidosis (DKA) in the 6 months prior to enrollment.
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 6 months prior to enrollment.
3. Current treatment of a seizure disorder.
4. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist.
5. Atrial or ventricular arrhythmias (benign premature atrial contractions [PACs] and premature ventricular contractions [PVCs] allowed)
6. Cystic fibrosis.
7. Pregnancy, breast-feeding, or intention of becoming pregnant over time of study procedures.
8. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

   i. Inpatient psychiatric treatment in the past 6 months ii. Presence of a known adrenal disorder iii. Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function iv. Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty v. Active gastroparesis vi. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study vii. Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise viii. Abuse of alcohol or recreational drugs ix. Infectious process not anticipated to be resolved prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis, deep tissue infection).

   x. Uncontrolled arterial hypertension (Resting diastolic blood pressure >100 mmHg and/or systolic blood pressure >180 mmHg).

   xi. Oral steroids xii. Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy) in the past 12 months.
9. A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol.
10. Basal Rates <0.01 units/hour for CSII subjects.
11. More than one basal dose per day for MDI subjects
12. Allergy for or intolerance of both Novolog (aspart) and Humalog (lispro) insulin for MDI subjects.
13. Diagnosed food allergies.
14. Current use of the following drugs and supplements:

    i. Regular acetaminophen user, or not willing to suspend acetaminophen 24 hours before and during the entire length of the trial ii. Any other medication that the investigator believes is a contraindication to the subject's participation
15. Any reason for which the study MD considers the subject not properly fitted for the trial (i.e. insulin pump that does not record what is needed for the trial).
16. Current enrollment in another clinical trial.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cherñavvsky, MD, CRC, Principal Investigator — UVA Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
To be determined

REFERENCES:
- [Result] Breton MD, Patek SD, Lv D, Schertz E, Robic J, Pinnata J, Kollar L, Barnett C, Wakeman C, Oliveri M, Fabris C, Chernavvsky D, Kovatchev BP, Anderson SM. Continuous Glucose Monitoring and Insulin Informed Advisory System with Automated Titration and Dosing of Insulin Reduces Glucose Variability in Type 1 Diabetes Mellitus. Diabetes Technol Ther. 2018 Aug;20(8):531-540. doi: 10.1089/dia.2018.0079. Epub 2018 Jul 6. PMID 29979618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-three subjects started the study. Nine discontinued after starting the study intervention: (1) data collection issues,(1) insulin parameter change needed, (5) personal reasons, and two subjects met stopping criteria - (1) glucagon & (1) high ketones; 24 subjects completed the protocol.
Pre-assignment Details: Blinded continuous glucose monitor (CGM) data will be collected for ~28 days prior to the Experimental Admission and analyzed by the study team to determine the optimal insulin therapy parameters for each insulin pump and multiple daily injections (MDI) participant. These optimized parameters will be used during the ~48 hour Experimental Admission.
Groups:
- Experimental (Decision Support) Admission, Then Control (Usual Care) Admission: Blinded CGM data was collected for ~28 days prior to the Experimental Admission & analyzed by the study team to determine the optimal insulin therapy parameters that would be used during the ~48 hour admission. Participants were instructed to record all meal information (i.e. carbohydrate quantity, insulin and self-monitoring blood glucose [SMBGs]) in the insulin pump during this Data Collection Phase.
  During the Experimental Admission, the DiAs (controlling the study pump) was programmed with the new optimized basal rates, correction factor, and carbohydrate ratios. These new parameters were applied during the entire admission. Once the insulin pump was functional, the pump dispensed insulin based on the optimized basal rates. The DiAs was "blinded", meaning the DiAs User Interface didn't display the CGM value, the DiAs plots, nor the amount of insulin dispensed. The admission was 48 hrs with controlled meals and exercise.
  During the Control Admission, the DiAs (controlling the study pump) was programmed with the subject's personnel parameters. The study subject determined the amount of insulin treatment during the admission. Subjects interacted with DiAs as a conventional bolus wizard. The admission was 48 hrs with controlled meals and exercise.
  The Experimental and Control Admission were separated by approximately 4 weeks, 8 weeks or 12 weeks.
- Control (Usual Care) Admission, Then Experimental (Decision Support) Admission: During the Control Admission, the DiAs (controlling the study pump) was programmed with the subject's personal parameters. The study subject determined the amount of insulin treatment during the admission. Subjects interacted with DiAs as a conventional bolus wizard. The admission was 48 hrs with controlled meals and exercise.
  Blinded CGM data was collected for ~28 days prior to the Experimental Admission & analyzed by the study team to determine the optimal insulin therapy parameters that would be used during the ~48 hour admission. Participants were instructed to record all meal information (i.e. carbohydrate quantity, insulin and self-monitoring blood glucose [SMBGs]) in the insulin pump during this Data Collection Phase.
  During the Experimental Admission, the DiAs (controlling the study pump) was programmed with the new optimized basal rates, correction factor, and carbohydrate ratios. These new parameters were applied during the entire admission. Once the insulin pump was functional, the pump dispensed insulin based on the optimized basal rates. The DiAs was "blinded", meaning the DiAs User Interface didn't display the CGM value, the DiAs plots, nor the amount of insulin dispensed. The admission was 48 hrs with controlled meals and exercise.
  The Experimental and Control Admission were separated by approximately 4 weeks, 8 weeks or 12 weeks.
Period: First Invention
Arm/Group | Experimental (Decision Support) Admission, Then Control (Usual Care) Admission | Control (Usual Care) Admission, Then Experimental (Decision Support) Admission
Started | 19 | 14
Completed | 14 | 12
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Data collection issues | 1 | 0
Not completed — Stopping criteria | 0 | 1
Not completed — Changed parameters during trial | 1 | 0
Period: Second Intervention
Arm/Group | Experimental (Decision Support) Admission, Then Control (Usual Care) Admission | Control (Usual Care) Admission, Then Experimental (Decision Support) Admission
Started | 14 | 12
Completed | 12 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Stopping Criteria | 1 | 0
Period: Third Intervention
Arm/Group | Experimental (Decision Support) Admission, Then Control (Usual Care) Admission | Control (Usual Care) Admission, Then Experimental (Decision Support) Admission
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline characteristics of all study participants regardless of randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Type 1 Diabetes Mellitus (T1DM) duration [Mean (Standard Deviation); unit: years] | 21 (11.1)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage] | 7.2 (1)
Height [Mean (Standard Deviation); unit: cm] | 172 (10.7)
Weight [Mean (Standard Deviation); unit: kg] | 81.8 (19.9)
Body Mass Index (BMI), kg/m2 [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (4.6)
Total Daily Insulin (TDI) [Mean (Standard Deviation); unit: U] | 46.7 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Glucose Variability (Coefficient of Variation)
Description: Assess effectiveness of glucose variability (GV) advisory system in reducing glucose variability in T1DM patient using an insulin pump.
Time Frame: Duration of the 48 hour study admission
Population: 24 participants completed the study. Data from subjects who withdrew were removed from analysis regardless of the degree of protocol completion.
Measure: Mean (Standard Deviation); unit: coefficient of variation
Groups:
- Decision Support System: Blinded CGM data was collected prior to the Experimental Admission and analyzed by the study team to determine the optimal insulin therapy parameters that was used during the Experimental Admission. The system was deployed on a portable medical application platform (DiAs) and include the following elements:
  1. An insulin pump treatment parameters optimization routine, using a month of collected CGM/insulin/meal data
  2. An exercise risk warning system, capable of predicting hypoglycemia at the onset of physical activity and advising on mitigating alteration of treatment.
- Usual Care (Control): Subjects used their own insulin parameters, including basal rate, correction factor and carbohydrate-insulin ratio, and determine their own insulin usage during the Control Admission.
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
coefficient of variation
  Overall | 0.33 (0.06) | 0.36 (0.08)
  Mealtime (4h following lunch and dinner) | 0.3 (0.07) | 0.34 (0.09)
  Overnight (11 pm-7 am) | 0.25 (0.08) | 0.28 (0.1)
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); Primary statistical analysis was performed using the repeated measure ANOVA, with the treatment mode as within subject factor, and type of insulin treatment (pump vs. MDI) as between subject factor. Based on achieved recruitment, a moderate effect size (0.3) is detectable with 80% power, or a large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for overall; Test type: Other; p = 0.045, ANOVA — No a priori sample size was determined due to the feasibility/pilot nature of the trial. Significance level was set at P-value <0.05
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); Primary statistical analysis was performed using the repeated measure ANOVA, with the treatment mode as within subject factor, and type of insulin treatment (pump vs. MDI) as between subject factor. Based on achieved recruitment, a moderate effect size (0.3) is detectable with 80% power, or a large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for mealtime; Test type: Other; p = 0.07, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); Primary statistical analysis was performed using the repeated measure ANOVA, with the treatment mode as within subject factor, and type of insulin treatment (pump vs. MDI) as between subject factor. Based on achieved recruitment, a moderate effect size (0.3) is detectable with 80% power, or a large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for overnight; Test type: Other; p = 0.177, ANOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Low Blood Glucose Index (LBGI)
Description: Low blood glucose index (LBGI) by CGM with higher index indicating higher risk of hypoglycemia. Values <1 suggest minimal risk. Index of risk of low blood glucose excursion based on a standard formula for non-linear transformation of the blood glucose scale (Kovatchev BP, Cox DJ, Gonder-Frederick LA, Young-Hyman D, Schlundt D, Clarke WL: Assessment of risk for severe hypoglycemia among adults with IDDM (Insulin dependent diabetes mellitus): validation of the low blood glucose index. Diabetes Care 21:1870-1875, 1998)
Time Frame: 48 hour study admission, outcomes were further divided into segments of the day: overnight (11 pm- 7 am).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LBGI
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
LBGI
  Overall | 1.59 (1.27) | 2.49 (2.08)
  Overnight | 1.89 (1.83) | 2.18 (1.96)
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); Secondary analysis followed the same format unless variables could not be considered normally distributed; in that case a related samples Wilcoxon signed-rank test was used. Data were first binned (to ensure minimum count of five per bins) & w2 statistics was used with expected counts given by standard of care. Based on achieved recruitment, moderate effect size (0.3) was detectable with 80% power, or large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for overall; Test type: Other; p = 0.042, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); Secondary analysis followed the same format unless variables could not be considered normally distributed; in that case a related samples Wilcoxon signed-rank test is used. Data were first binned (to ensure minimum count of five per bins) and the w2 statistics was used with the expected counts given by SoC. Based on achieved recruitment, a moderate effect size (0.3) is detectable with 80% power, or a large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for overnight; Test type: Other; p = 0.276, ANOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Below 50 mg/dL
Description: CGM measured blood sugar values below 50 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 50 mg/dL is considered a better outcome.
Time Frame: 48 hour study admission, outcomes were further divided into segments of the day: overnight (11 pm- 7 am), and around meals (the 4 h following lunch and dinner, breakfast excluded due to exercise).
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 0 [0 to 0] | 0 [0 to 0.7]
  Mealtime | 0 [0 to 0] | 0 [0 to 0]
  Overnight | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); Secondary analysis followed the same format unless variables could not be considered normally distributed; in that case a related samples Wilcoxon signed-rank test is used. Data were first binned (to ensure minimum count of five per bins) and the w2 statistics was used with the expected counts given by SoC. Based on achieved recruitment, a moderate effect size (0.3) is detectable with 80% power, or a large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for overall; Test type: Other; p = 0.026, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); Secondary analysis followed the same format unless variables could not be considered normally distributed; in that case a related samples Wilcoxon signed-rank test is used. Data were first binned (to ensure minimum count of five per bins) and the w2 statistics was used with the expected counts given by SoC. Based on achieved recruitment, a moderate effect size (0.3) is detectable with 80% power, or a large effect size (0.4) with 95% power (G-Power 3.1.9.2). Outcome measurement was for mealtime; Test type: Other; p = 0.173, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.715, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Below 60 mg/dL
Description: CGM measured blood sugar values below 60 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 60 mg/dL is considered a better outcome.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 0.1 [0 to 0.5] | 0.66 [0 to 1.6]
  Mealtime | 0 [0 to 0.4] | 0 [0 to 1.7]
  Overnight | 0 [0 to 0.3] | 0 [0 to 1.9]
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.036, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.213, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.110, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percent Below 70 mg/dL
Description: CGM measured blood sugar values below 70 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 70 mg/dL is considered a better outcome.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 0.88 [0.4 to 2.3] | 3.21 [1.3 to 4.8]
  Mealtime | 1.23 [0 to 3.2] | 1.73 [0.5 to 5.2]
  Overnight | 1.15 [0 to 3.2] | 3.33 [0 to 5.6]
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.018, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.149, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.109, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percent Between 70 and 180 mg/dL
Description: CGM measured blood sugar values between 70 abd 180 mg/dL are considered to be desirable. A higher percentage of time in this range is indicative of a desirable outcome.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 68.9 (14.3) | 65.9 (18.6)
  Mealtime | 77.9 (19.2) | 73.3 (27.3)
  Overnight | 68.2 (20.3) | 63 (23.5)
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.78, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.399, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.824, ANOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percent Above 180 mg/dL
Description: CGM measured blood sugar values above 180 mg/dL are considered to be undesirable. Thus, less time spent above 180 mg/dL is considered a positive outcome
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 29.4 (15.6) | 30.3 (19.5)
  Mealtime | 19.9 (20.4) | 23.6 (27.9)
  Overnight | 29.2 (21.7) | 31.2 (25)
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.863, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.965, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.742, ANOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percent Above 250 mg/dL
Description: CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250 mg/dL is considered a positive outcome
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 5.2 [0 to 11.5] | 6.3 [3.5 to 14.7]
  Mealtime | 0 [0 to 0.1] | 0 [0 to 8.9]
  Overnight | 0 [0 to 8.6] | 7.4 [0 to 15.9]
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.158, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.085, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.055, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percent Above 300 mg/dL
Description: CGM measured blood sugar values above 300 mg/dL are considered to be undesirable. Thus, less time spent above 300 mg/dL is considered a positive outcome
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
percentage of time
  Overall | 0 [0 to 4.5] | 1 [0 to 2.6]
  Mealtime | 0 [0 to 0] | 0 [0 to 0]
  Overnight | 0 [0 to 0] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.744, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.248, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.225, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Average Glycemia (mg/dL)
Description: Average glycemia is a measure of the average CGM value in mg/dL during the 48 hour study admission. A lower value, without approaching hypoglycemia, is indicative of a desirable outcome.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
mg/dL
  Overall | 155.2 (23.2) | 155.2 (27.1)
  Mealtime | 142.7 (29.7) | 144 (35.5)
  Overnight | 151.9 (29.9) | 156.9 (37.6)
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.86, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 2]; Test type: Other; p = 0.522, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 2, analysis 2]; Test type: Other; p = 0.522, ANOVA — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Total Insulin Used
Description: This measure is an average of the total amount of insulin (both basal and bolus) used by participants during the study admission.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U
Arm/Group | Decision Support System | Usual Care (Control)
Number analyzed (Participants) | 24 | 24
U | 44.1 (18.4) | 45.5 (22.8)
Statistical Analysis 1: Comparison: Decision Support System vs Usual Care (Control); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.301, ANOVA — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Basal Insulin Used
Description: This measure is an average of the total amount of basal insulin used by participants during the study admission.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U
Groups:
- Control (Usual Care) Admission, Data Collection, Then Experimental (Decision Support) Admission: Subjects used their own insulin parameters, including basal rate, correction factor and carbohydrate-insulin ratio, and determine their own insulin usage during the Control Admission.
  Blinded CGM data was collected prior to the Experimental Admission and analyzed by the study team to determine the optimal insulin therapy parameters that was used during the Experimental Admission.
  Decision Support System: The purpose of this study was to demonstrate the safety and feasibility of a Decision Support System aimed at reducing glucose variability in T1DM patient using an insulin pump. The system was deployed on a portable medical application platform (DiAs) and include the following elements:
  1. An insulin pump treatment parameters optimization routine, using a month of collected CGM/insulin/meal data
  2. An exercise risk warning system, capable of predicting hypoglycemia at the onset of physical activity and advising on mitigating alteration of treatment.
Arm/Group | Decision Support System | Control (Usual Care) Admission, Data Collection, Then Experimental (Decision Support) Admission
Number analyzed (Participants) | 24 | 24
U | 20.3 (9.1) | 21.4 (11.1)
Statistical Analysis 1: Comparison: Decision Support System vs Control (Usual Care) Admission, Data Collection, Then Experimental (Decision Support) Admission; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.189, ANOVA — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Total Rescue Carbohydrates (CHO) (Grams)
Description: The average of the total amount of rescue carbohydrates (grams) administered during the study admission under safety protocols. Administering fewer carbohydrates is a desirable outcome because it indicates better control.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Decision Support System | Control (Usual Care) Admission, Data Collection, Then Experimental (Decision Support) Admission
Number analyzed (Participants) | 24 | 24
g | 81 (74.2) | 96 (78.1)
Statistical Analysis 1: Comparison: Decision Support System vs Control (Usual Care) Admission, Data Collection, Then Experimental (Decision Support) Admission; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.271, ANOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately 10 weeks
Groups:
- Decision Support System: Blinded CGM data will be collected prior to the Experimental Admission and analyzed by the study team to determine the optimal insulin therapy parameters that will be used during the Experimental Admission.
  Decision Support System: The purpose of this study is to demonstrate the safety and feasibility of a Decision Support System aimed at reducing glucose variability in T1DM patient using an insulin pump. The system will be deployed on our portable medical application platform (DiAs) and will include the following elements:
  1. An insulin pump treatment parameters optimization routine, using a month of collected CGM/insulin/meal data
  2. An exercise risk warning system, capable of predicting hypoglycemia at the onset of physical activity and advising on mitigating alteration of treatment.
- Usual Care: Subjects will use their own insulin parameters, including basal rate, correction factor and carbohydrate-insulin ratio, and determine their own insulin usage during the Control Admission.
Arm/Group | Decision Support System | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 1/33 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decision Support System (N=33) | Usual Care (N=33)
Hypoglycemia requiring glucagon administration (Endocrine disorders) | 0 (0) | 1 (1) — Did extreme exercise. Administered meal insulin/blood glucose (BG)=~50s. Treated with fast acting carbs 3 times as BG continued to drop. Self-administered glucagon to stabilize BG. Dropped from study - didn't complete Exp study so data not used.
Ketones (Endocrine disorders) | 1 (1) | 0 (0)
Respiratory illness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Herpetic Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bump on head (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT02558491/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT02558491/ICF_001.pdf